CLINICAL TRIAL: NCT06603428
Title: Functional Outcome in Operative and Nonoperative Management in Isolated Greater Tuberosity Fracture of Humerus Bone: (cohort Study)
Brief Title: Functional Outcome in Operative and Nonoperative Management in Isolated Greater Tuberosity Fracture of Humerus Bone
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Kerollos Zaghloul Thabet, asisstant lecturer, Assiut University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: greater tuberosity fracture
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Greater Tuberosity Fracture
MeSH Terms: conditions — Shoulder Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Operative and Nonoperative Management in Isolated Greater Tuberosity Fracture of Humerus Bone. (Experimental): Patients more than 5 ml displacement of GT fracture (3ml in active highly demanded patient) are for internal fixation, others less this are for conservative management.
  Interventions: Device: internal fixation by plate or screws

INTERVENTIONS:
Device: internal fixation by plate or screws — - Patients more than 5 ml displacement of GT fracture (3ml in active highly demanded patient) are for internal fixation, others less this are for conservative management.
  Other Names: arthroscopic fixation of avulsion greater tuberosity fracture

SUMMARY:
Constant score for functional outcome in operative and non-operative management in isolated greater tuberosity fractures of humerus bone.

DETAILED DESCRIPTION:
Fractures of the greater tuberosity (GT) often occur with more complex proximal humerus fractures and are less frequently observed as an isolated pathology. Only 14-20% of proximal humerus fractures are isolated lesions of the GT. Up to 30% of these fractures are associated with anterior glenohumeral dislocations. According to Neer, a displacement of the fragment >5mm and 30°, or >3 mm of displacement in active patients involved in frequent overhead activity is believed to be an indication for operative treatment. However, indication for all other fractures had managed by nonoperative treatment is unclear. Currently, there is a lack of evidence in the literature to support either conservative or operative treatment strategies in GT humerus fractures. The fracture type and the etiology of the fracture impact the decision- making and the final outcome also remains unclear. age of more than 65 years as an important risk factor for secondary displacement in the conservative management of fractures of the greater tuberosity. Furthermore, fracture type and shoulder joint dislocations were factors associated with show increased relative risks for secondary fragment displacement.

ELIGIBILITY:
Inclusion Criteria:

* 1-history of traumatic isolated GT fracture.

Exclusion Criteria:

- 1- associated proximal humeral fracture.

2 - previous shoulder pathology.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-10-10 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Constant score for functional outcomes | follow up 1 year
  A-Pain (/15): Average(1+2) A
  1. Do you have pain in your shoulder (normal activities)? No =15 pts,Mild pain =10 pts,Moderate =5 pts,Severe or permanent =0.
  2. Linear scale:
  If "0" means no pain and "15" is the maximum pain you can experience, please circle where is the level of pain of your shoulder.(Points given are inverse to the scale.E.g. level 5 in the scale means 10 points) B- Activities of daily living (/20) Total (1 + 2) B
  1. Is your occupation or daily living limited by your shoulder? No=4,Moderate limitation =2,Severe limitation=0
  2. Are your leisure and recreational activities limited by your shoulder? No=4,Moderate limitation = 2,Severe limitation=0 C.- Range of movement (leave this for the doctor or physiotherapist) (/40):Total (1 + 2 ) C
  1.- FWD Flexion: 0-30 0 pts 2-Abduction: 0-30 D.- Power (/25): Points: average (kg) x 2= D
  First pull:Second pull:Third pull:Fourth pull:Fifth pull:
  Average pulls:
  TOTA

CONTACTS AND LOCATIONS:
Overall Officials: Kerolos Z Thabet, master, Principal Investigator — Assiut University
Locations (1):
- Kerolos Zaghlol Thabet, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
For conservative cases
  * 1ist 4 weeks abduction sling.
  * 2end 2 weeks active assisted movement + abduction sling.
  * After 6 weeks active movement. For operative cases
  * Day one passive movement.
  * After 4 weeks active assisted movement.
  * After 6 weeks active movement
Supporting Information: Study Protocol, SAP
Time Frame: Follow up conservative and operative cases for one year, radiological assessment by x-ray and clinical assessment follow up at 1.5,3,6,9 month and at 1 year using Constant score
Access Criteria: 1. isolated GT fracture
  2. age 20-60

REFERENCES:
- [Background] Schliemann B, Heilmann LF, Raschke MJ, Lill H, Katthagen JC, Ellwein A. Isolated fractures of the greater tuberosity: When are they treated conservatively?: A baseline study. Obere Extrem. 2018;13(2):106-111. doi: 10.1007/s11678-018-0459-z. Epub 2018 May 15. PMID 29887916